CLINICAL TRIAL: NCT05242237
Title: The Prognostic Value of Circulating Tumor Cells Isolated by a Novel Microfluidic Platform in Liver Cancer Patients
Brief Title: Prognostic Value of Liver Cancer CTCs Isolated by a Novel Microfluidic Platform
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Second Affiliated Hospital of Chongqing Medical University (Other)
Collaborators: Cellomics International Limited (Unknown)
Responsible Party: Principal Investigator, Zhihang Zhou, Professor, The Second Affiliated Hospital of Chongqing Medical University
Other Study IDs: HCC-CTC
Record Dates: First submitted 2022-01-24; First posted 2022-02-16 (Actual); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: Hepatocellular Carcinoma; Circulating Tumor Cell; Whole Genome Sequencing
Keywords: whole genome sequencing; microfluidic device; inertial focus
MeSH Terms: conditions — Carcinoma, Hepatocellular; Neoplastic Cells, Circulating

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HCC patients: HCC patients with initial diagnosis
- Liver cirrhosis patients: Liver cirrhosis patients

SUMMARY:
This study aims to isolate CTCs in peripheral venous blood of liver cancer patients by inertial focusing principle-based microfluidic device, determine the relationship between the number of CTCs and patient prognosis and treatment response, detect mutation, copy number variation and mutation load in CTC cells and corresponding tissues using single-cell whole genome sequencing technology, and use bioinformatics analysis of CTC heterogeneity and its relationship with clinical outcome. In addition, the culture of CTCs in vitro was explored by organoid culture or sphere culture in order to obtain CTCs cell lines to reveal the metastatic mechanisms of HCC. The partner of this project is Cellomics International Limited, which could provide Cellomics CTC-100 cell sorter and related consumables for this project. Peripheral venous blood from about 300 patients with initial liver cancer will be collected, and CTCs cells will be sorted in 8ml of each patient and typed according to protein expression. Clinical data, treatment effect and survival time of patients will be collected, and finally the relationship between the number of CTCs and subgroup with treatment response and patient prognosis will be analyzed. Uncovering the genomic characteristics of CTCs of HCC provides a new basis for the precise treatment of HCC. The new diagnostic markers for Hcancer were found by miRNA expression spectrum chip and metabolomic testing.In vitro culture methods and cellular characteristics of HCC circulating tumor cells were preliminarily explored.

DETAILED DESCRIPTION:
In China, the incidence of hepatocellular carcinoma (HCC) ranks the fourth, and the mortality rate is the second. Less than 20% of the patients were able to receive curative resection therapy. Most other patients with HCC have a very poor prognosis, with only chemical embolization, ablation treatment or systemic treatment, and the treatment effect is limited. Effective markers are required for the early diagnosis, treatment, prediction of prognosis, and assessment of treatment response in HCC. At present, alpha-fetoprotein (AFP) is the most common marker of HCC, which can be used for its diagnosis and patient prognosis. However, AFP has less sensitivity in the diagnosis of HCC. Although some other markers, such as AFP heteromer, abnormal prothrombin, also have a role in the diagnosis of HCC, they have not been widely used in clinical practice. Liver biopsy helps to directly evaluate the molecular biology of the tumor, but it has the risk of bleeding and causing tumor dissemination, which is currently rarely used in the diagnosis of HCC. Furthermore, liver puncture biopsy due to tumor heterogeneity may not adequately reflect the overall tumor characteristic.

Liquid biopsy can be used in various aspects of tumor diagnosis, detection and treatment, including circulating tumor cells, circulating tumor DNA, circulating miRNA, metabolites, etc. Circulating tumor cells (circulating tumor cells, CTCs) from the tumor group into the circulating system of tumor cells, is the key factor of tumor metastasis. Most CTCs can die from anoikisis, immune attack, or shear stress. To adapt to the environment, CTCs undergo a range of changes, such as epithelial-mesenchymal transition (EMT). Tumor cells undergo EMT and lose epithelial cell markers and acquire stromal cell features. Thus, CTCs are a group of cells derived from different regions of tumor tissue that are heterogeneous and play a critical role in tumor progression. CTCs are not only minimally invasive, but also can reflect the heterogeneity of tumor tissue. The CTCs convey the genomic information from the primary tumor tissue, which can indirectly reflect the information about the gene mutation, the copy number variation, and the tumor mutation load in the tumor tissue through the whole-genome sequencing of the CTCs, helping the clinicians to develop the treatment plan. For example, preliminary studies have shown that copy number variation in CTCs has a high accordance with primary HCC tissues.

CTCs have been extensively studied in multiple solid tumors. For example, in patients with metastatic prostate cancer, the number of CTCs can accurately predict the prognosis of the patients and reflect the of the treatment. Examination HER2-positive CTCs cells in breast cancer patients helps to specify the designated patient's treatment regimen. However, in patients with HCC surgical resection, the number of CTC was associated with of vascular invasion, AFP level, tumor stage, tumor progression, and patient poor prognosis. Recently, it has been shown that postoperative adjuvant TACE is able to prolong the survival time of patients after HCC resection with preoperative EpCAM-positive CTC, with no significant effect on in CTC-negative patients. However, the number of CTCs was minimal, and the heterogeneity existed. There are many limitations on the detection of CTCs, and how to accurately detect CTCs is still a problem that bothers us. The presently used platform for isolating CTCs is based primarily on tumor cell markers, biophysical properties, or strategies without enrichment. Isolation based on tumor surface markers was sorted using specific antibodies: leukocytes were removed from leukocyte surface markers (such as CD45), that is, negative sorting; CTCs were separated from tumor cell surface markers (EpCAM, ASGPR, CK), i. e., positive sorting. The limitation of this approach is the fact that selection of markers fails to reflect tumor heterogeneity and reduces cellular activity. Separation methods based on the cell volume, elasticity, and conductance of CTCs, such as microfiltration, gradient centrifugation, and inertial focus, avoid the limitations of using surface markers for separation while having little effect on cell activity. Without enrichment methods, using high-speed fluorescence imaging, can distinguish CTCs directly in patients' blood.

The CTC-100 circulating tumor cell detection system used by Shenzhen Jingyi Medical Laboratory has been filed for the record of Shenzhen Class I medical devices (record No.: No.20190047) and has been on the market. The system is capable of efficiently capturing the enriched CTC. It mainly relies on the inertial focusing principle of the microfluidic chip and the elastic physical characteristics to realize the screening. This device makes the fluid laminar in the straight channel, the fluid near the channel wall is lowest, while the maximum fluid velocity in the middle of the channel. This flow velocity distribution produces a shear force gradient, and induces the resulting lift will push the particles to the wall. When it moves close to the wall of the channel, the lift induced by the channel wall again pushes the particles away from the channel wall. Both lift forces in opposite directions are called inertial lift, this force acts on the particles, moves it to the equilibrium position. Thus the particles focus on the stable site, form a focused flow. Cell particles migrate with liquid migration in microfluidic chip channels, due to the different size and elasticity of CTC and white blood cells, finally focusing on different equilibrium positions, thus achieving the screening effect. Screened tumor cells can identify their surface glycochemical characteristics and biological characteristics (EpCAM, PDL1, VEGF, etc.), and finally achieve high sensitivity and specific CTC screening and identification. Our preclinical trials showed that the number of CTC tested by this technique was significantly higher in liver cancer patients than in cirrhosis and healthy patients, and was positively associated with liver vascular invasion and tumor size (102 liver cancer, 43 cirrhosis and 10 healthy patients). The detection rate of this technique was 100% in HCC patients, and 64.7% of the cells detected in the CTC were EpCAM negative.Whole-genome sequencing found that the gene mutations in the CTC were consistent with the corresponding cancer tissue (5 CTC samples and the corresponding surgical resection tissue), suggesting that the CTCs can reflect information such as gene mutations in the cancer tissue.

This study aims to isolate CTCs in peripheral venous blood of liver cancer patients by inertial focusing principle-based microfluidic device, determine the relationship between the number of CTCs and patient prognosis and treatment response, detect mutation, copy number variation and mutation load in CTC cells and corresponding tissues using single-cell whole genome sequencing technology, and use bioinformatics analysis of CTC heterogeneity and its relationship with clinical outcome. In addition, the culture of CTCs in vitro was explored by organoid culture or sphere culture in order to obtain CTCs cell lines to reveal the metastatic mechanisms of HCC. The partner of this project is Cellomics International Limited, which could provide Cellomics CTC-100 cell sorter and related consumables for this project. Peripheral venous blood from about 300 patients with initial liver cancer will be collected, and CTCs cells will be sorted in 8ml of each patient and typed according to protein expression. Clinical data, treatment effect and survival time of patients will be collected, and finally the relationship between the number of CTCs and subgroup with treatment response and patient prognosis will be analyzed. Uncovering the genomic characteristics of CTCs of HCC provides a new basis for the precise treatment of HCC. The new diagnostic markers for Hcancer were found by miRNA expression spectrum chip and metabolomic testing.In vitro culture methods and cellular characteristics of HCC circulating tumor cells were preliminarily explored.

ELIGIBILITY:
Inclusion Criteria:

* confirmed by imaging and serological examination for benign liver cancer;
* patients without any previous treatment;
* informed consent;
* age: 18 years or older (adult).

Exclusion Criteria:

* with other malignancies;
* metastatic liver tumors;
* with major organic lesions;
* with acute complications such as acute liver failure, massive gastrointestinal bleeding and so on.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Peripheral venous blood samples are expected to collect 300 liver cancer patients and 50 patients with liver cirrhosis, taking 8ml of venous blood from each patient. Among them, about 100 patients underwent surgery (about 5 * 5 * 5mm).After receiving follow-up for 1-2 years, information on patient treatment regimen, treatment response, recurrence, metastasis, survival time and other patients was collected.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2024-01-31 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
Time to progression or death (months) | 2 years
  Time to progression or death (months) after initial diagnosis will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: ZHOU ZHIHANG, Principal Investigator — The Second Affiliated Hospital of Chongqing Medical University
Locations (1):
- the second affiliated hospital of Chongqing Medical University, Chongqing, China

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared after the trial has been finished
Supporting Information: Study Protocol, CSR
Time Frame: will be shared after the trial has been finished

REFERENCES:
- [Result] Llovet JM, Kelley RK, Villanueva A, Singal AG, Pikarsky E, Roayaie S, Lencioni R, Koike K, Zucman-Rossi J, Finn RS. Hepatocellular carcinoma. Nat Rev Dis Primers. 2021 Jan 21;7(1):6. doi: 10.1038/s41572-020-00240-3. PMID 33479224
- [Result] Ahn JC, Teng PC, Chen PJ, Posadas E, Tseng HR, Lu SC, Yang JD. Detection of Circulating Tumor Cells and Their Implications as a Biomarker for Diagnosis, Prognostication, and Therapeutic Monitoring in Hepatocellular Carcinoma. Hepatology. 2021 Jan;73(1):422-436. doi: 10.1002/hep.31165. Epub 2021 Jan 18. PMID 32017145
- [Result] Chen VL, Xu D, Wicha MS, Lok AS, Parikh ND. Utility of Liquid Biopsy Analysis in Detection of Hepatocellular Carcinoma, Determination of Prognosis, and Disease Monitoring: A Systematic Review. Clin Gastroenterol Hepatol. 2020 Dec;18(13):2879-2902.e9. doi: 10.1016/j.cgh.2020.04.019. Epub 2020 Apr 11. PMID 32289533
- [Result] Zhu Z, Qiu S, Shao K, Hou Y. Progress and challenges of sequencing and analyzing circulating tumor cells. Cell Biol Toxicol. 2018 Oct;34(5):405-415. doi: 10.1007/s10565-017-9418-5. Epub 2017 Nov 22. PMID 29168077
- [Result] Court CM, Hou S, Liu L, Winograd P, DiPardo BJ, Liu SX, Chen PJ, Zhu Y, Smalley M, Zhang R, Sadeghi S, Finn RS, Kaldas FM, Busuttil RW, Zhou XJ, Tseng HR, Tomlinson JS, Graeber TG, Agopian VG. Somatic copy number profiling from hepatocellular carcinoma circulating tumor cells. NPJ Precis Oncol. 2020 Jul 2;4:16. doi: 10.1038/s41698-020-0123-0. eCollection 2020. PMID 32637655
- [Result] Pantel K, Hille C, Scher HI. Circulating Tumor Cells in Prostate Cancer: From Discovery to Clinical Utility. Clin Chem. 2019 Jan;65(1):87-99. doi: 10.1373/clinchem.2018.287102. PMID 30602476
- [Result] Chen W, Zhang J, Huang L, Chen L, Zhou Y, Tang D, Xie Y, Wang H, Huang C. Detection of HER2-positive Circulating Tumor Cells Using the LiquidBiopsy System in Breast Cancer. Clin Breast Cancer. 2019 Feb;19(1):e239-e246. doi: 10.1016/j.clbc.2018.10.009. Epub 2018 Nov 1. PMID 30472074
- [Result] Wang PX, Sun YF, Zhou KQ, Cheng JW, Hu B, Guo W, Yin Y, Huang JF, Zhou J, Fan J, Cheung TT, Qu XD, Yang XR. Circulating tumor cells are an indicator for the administration of adjuvant transarterial chemoembolization in hepatocellular carcinoma: A single-center, retrospective, propensity-matched study. Clin Transl Med. 2020 Jul;10(3):e137. doi: 10.1002/ctm2.137. Epub 2020 Jul 23. PMID 32702202
- [Result] Jackson JM, Witek MA, Kamande JW, Soper SA. Materials and microfluidics: enabling the efficient isolation and analysis of circulating tumour cells. Chem Soc Rev. 2017 Jul 17;46(14):4245-4280. doi: 10.1039/c7cs00016b. PMID 28632258